CLINICAL TRIAL: NCT00732719
Title: A Phase II Non-Comparative Study Evaluating the Effects of the Compression Test Device on Oedema
Brief Title: Compression Device Safety Study on Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Professor Wolfgang Vanscheidt, Hautarzt Phlebologe Allergologe
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CW-0500-04-U332
Record Dates: First submitted 2008-07-23; First posted 2008-08-12 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-08

CONDITIONS: Edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Profile A (Placebo Comparator): Device worn; no pressure given (placebo)
  Interventions: Device: Prototype device (unnamed) worn-no pressure given (placebo) from inflatable cuffs
- Profile B (Active Comparator): Foot at 30mm Hg, Gaiter at 40 mm Hg, mid-calf at 30 mm Hg and upper cuff at 20mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile C (Active Comparator): Foot at 20mm Hg, Gaiter at 30 mm Hg, mid-calf at 20 mm Hg and upper cuff at 10mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile D (Active Comparator): Foot at 10mm Hg, Gaiter at 20 mm Hg, mid-calf at 10 mm Hg and upper cuff at 0mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile E (Active Comparator): Foot at 30mm Hg, Gaiter at 40 mm Hg, mid-calf at 40 mm Hg and upper cuff at 40mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile F (Active Comparator): Foot at 20mm Hg, Gaiter at 30 mm Hg, mid-calf at 30 mm Hg and upper cuff at 30mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile G (Active Comparator): Foot at 10mm Hg, Gaiter at 20 mm Hg, mid-calf at 20 mm Hg and upper cuff at 20mm Hg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs

INTERVENTIONS:
Device: Prototype device (unnamed) worn-no pressure given (placebo) from inflatable cuffs
  Arms: Profile A
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile B
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile C
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile D
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile E
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile F
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile G

SUMMARY:
To evaluate the safety of the prototype Compression Device in subjects with Oedema

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 80, willing and able to provide written informed consent, and able to wear the device and follow the requirements of the protocol
* Subjects who have an ankle to brachial pressure index (ABPI) of at least 0.8.
* Subjects who suffer from chronic oedema (i.e. CEAP classification of C3, C4 or C5 1.)
* Subjects who have Chronic Venous Insufficiency (CVI), which has been present for 6 weeks or longer and who have refluxes >0.5 sec in one or more major venous segments, superficial or deep or both (CEAP classification: C3-C5 1.; Ep,s; As,d; Pr).

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product.
* Subjects who have previously been entered into the study before
* Subjects who have a history of Deep Vein Thrombosis (DVT) within the last 6 months
* Subjects who have an active leg ulcer (i.e. CEAP classification of C6 1).
* Subjects with active cardiac disease or significant history of cardiac disease (including history of myocardial infarction, heart failure, valvular disease, arrhythmia and those with a pacemaker or have previously had a pacemaker).
* Subjects who have initiated treatment or changed the dose within the past month of pharmaceutical agents that reduce clotting e.g. aspirin (except low-dose aspirin), anti-platelets, anti-coagulants and coumarin.
* Subjects who are currently taking pharmaceutical agents that can modify the amount of leg oedema (e.g., diuretics, dihydropyridine calcium channel blockers, phlebotonic drugs, or fluctuating doses of systemic steroids) or have taken these agents within the last 10 days.
* Subjects who are pregnant
* Subjects who have worn compression therapy in the last 48 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The nature and incidence of adverse events
Volume reduction
Oedema reduction

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Vanscheidt, Principal Investigator — Hautarzt Phlebologe Allergologe
Locations (1):
- Hautarzt Phlebologe Allergologe, Freiburg im Breisgau, Germany